CLINICAL TRIAL: NCT06032780
Title: Effects of Eccentric Resistance Training on Ventricle Functions and Aerobic Capacity Among Individuals With Chronic Heart Failure
Brief Title: Eccentric Resistance Training Among Individuals With Chronic Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ISB/REC/PhD/01199 Iqbal Tariq
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Group allocation will be kept blinded to the assessor and to the treatment provider (trained physical therapist).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eccentric Resistive Training + Aerobic training Group (Experimental)
  Interventions: Other: Eccentric Resistive Training + Aerobic training Group
- Resistance Training + Aerobic training Group (Active Comparator)
  Interventions: Other: Resistance Training + Aerobic training Group
- Aerobic training Group (Active Comparator)
  Interventions: Other: Aerobic training Group

INTERVENTIONS:
Other: Eccentric Resistive Training + Aerobic training Group — Eccentric Resistive training includes upper limb (biceps and triceps) and lower limb large muscle training (quadriceps and hamstrings) 2 sets of 12 repetitions (reps) for each group of muscles in lengthened position for eccentric training in approx. 20 minutes (min). Intensity will be based on 1 repetition maximum (1RM) starting from 20% of (1RM) and its intensity in percentage will be progress by 10% after every two weeks. Stair descending training and squatting position and eccentric hamstring curls with weights at ankle for lower limb eccentric training progressive as per tolerance in response to modified Borg scale (with cut off of showing dyspnea of 4 somewhat hard) and Numeric Pain rating scale (with cut off of showing 7 on scale, crossing moderate pain) . (approx. 20 min).
  + Aerobic training as a control will be given to this group as well for approximately 30 minutes per session.
  Arms: Eccentric Resistive Training + Aerobic training Group
Other: Resistance Training + Aerobic training Group — Resistive training (concentric) includes Upper limb (biceps and triceps) and lower limb large muscle training (quadriceps and hamstrings), 2 sets of 12 reps for each group of muscles in approx. 30 min. Intensity will be based on 1 repetition maximum (1RM) starting from 20% of (1RM) and its intensity in percentage will be progress by 10% after every two weeks. Stair climbing training and quadriceps training + standing hamstring curls with weight at ankle for lower limb concentric training progressive as per tolerance in response to modified Borg scale (with cut off of showing dyspnea of 4 somewhat hard) and Numeric Pain rating scale (with cut off of showing 7 on scale, crossing moderate pain)
  + Aerobic training as a control will be given to this group as well for approximately 30 minutes per session.
  Arms: Resistance Training + Aerobic training Group
Other: Aerobic training Group — Aerobic training as a control will be given to this group as well for approximately 60 minutes per session. Aerobic training exercise will be completed via a ergometer/stationary cycle; type will be continuous aerobic exercise and intensity of 60% of max HR (or peak VO2) in HF individuals.
  Arms: Aerobic training Group

SUMMARY:
To determine the effects of eccentric resistive training on ventricle functions and aerobic capacity as compared to a resistance and aerobic training among Heart failure (HF)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic HF and currently stable with optimal medical therapy
* Chronic Heart failure with ejection fraction > 30 %
* Patient able to safely perform lower limb exercise will be check by six- minute walk test (6 MWT)

Exclusion Criteria:

* Those Heart failure patient whose are in acute phase or planed for any immediate medical intervention
* Already participating in cardiac rehabilitation
* New York Heart Association (NYHA) Classification of HF class IV HF symptoms
* Co-existent other disease such as asthma/ COPD/interstitial lung disease.
* Symptomatic Second degree or third degree heart block.
* ECG with uncontrolled ventricular arrhythmia
* Limited Exercise ability due to neurologic or orthopedic impairments of the legs (will cross-check with 6 MWT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Ventricle Functions | 12 week
  Changes from the baseline will be measured. Doppler resting echocardiography will be performed to measure ventricle functions. Standard views, including the parasternal long-axis, short-axis at the papillary muscle level, and apical 4- and 2-chamber views will be recorded. Left ventricular ejection fraction (LVEF) and end systolic and end-diastolic diameters (LVESD and LVEDD) will be measured using formula (Tiecholz formula i-e spherical volume of the heart multiplied by a correction factor). Any structural changes will also be recorded.
Aerobic Capacity | 12 week
  Changes will be measured at baseline, 4th week, 8th week and 12th week. The 6-min walk test provides an indirect measure of cardiovascular functional/aerobic capacity. Six Minute Walk test (6MWT) will be used to assess the functional capacity of the individuals with HF. The subjects will be instructed to walk for 6 minutes at a given time along a 30-m line at an interval of 1.5 m in an outdoor corridor, and the distance walked will be recorded in meters. The participants will be encouraged to continue walking as fast as possible. Then a generalized equation will be used to predict peak VO2 from 6 minute walk distance (6MWD) with the help of formula. Mean Peak VO2 (ml/kg/Mean) = 4.948 + 0.023 *Mean 6MWD (meters)

SECONDARY OUTCOMES:
Quality of life (Minnesota Living with Heart Failure Questionnaire) | 12 week
  Changes from the baseline will be measured. Quality of life will be measured through Minnesota Living with Heart Failure Questionnaire (MLHFQ). It is one of the most widely used health-related quality of life questionnaires for individuals with HF. It provides scores for two dimensions, physical and emotional, and a total score. The MLHFQ is a self-administered, 21-item disease-specific instrument for individuals with HF. Each item is scored in a 6-point Likert Scale (0 to 5), thus the total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life. The MLHFQ has two domains; physical domain (eight items, score range from 0 to 40) and emotional domain (five items, score range from 0 to 25).
Strength | 12 week
  Changes will be measured at baseline, 4th week, 8th week and 12th week. Maximum muscle strength of the all major muscles biceps, triceps, quadriceps and hamstring, will be measured in sitting position with (MicroFET2 Digital Handheld Dynamometer muscle tester).
Maximal strength of respiratory muscles | 12 week
  Changes will be measured at baseline, 4th week, 8th week and 12th week. Maximum Inspiratory pressure (MIP) and Maximal Expiratory pressure (MEP) will be assessed through a handheld mouth pressure meter.
Forced Expiratory Volume in 1 second (FEV1) | 12 week
  Changes will be measured at baseline, 4th week, 8th week and 12th week, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 12 week
  Changes will be measured at baseline, 4th week, 8th week and 12th week, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters
Peak Expiratory Flow (PEF) | 12 week
  Changes will be measured at baseline, 4th week, 8th week and 12th week, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second.
Cardiac Risk Factors - Blood Pressure | 12 week
  Changes from the Baseline, Blood pressure (Bp) (both systolic/diastolic) will be measured in mmHg. It will be measured manually through sphygmomanometer by trained assessor in sitting position at baseline and at end of training on each week (for safety check).
Cardiac Risk Factors - Body mass index | 12 week
  Changes will be measured at baseline, 6th week and at 12th week. Weight in kilograms (kg) and Height in meters (m) will be combined to report BMI in kg/m^2 to measure the Body mass index
Cardiac Risk Factors - Lipid profile | 12 week
  Changes form the baseline, The lipid profile includes total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), and triglyceride (TG). All units are in mmol/L.

OTHER OUTCOMES:
Oxygen Saturation (SpO2) | 12 week
  Changes from baseline SPO2 was measured in percentage. Oxygen immersion is the division of oxygen-soaked hemoglobin with respect to add up to hemoglobin in the blood. Pulse oximeter measure it. It will also be measured on each week (for safety check)
Change in heart rate variability (HRV) | 12 week
  HRV is obtained from the spectral analysis of R-R intervals obtained from a heart rate monitor (Polar belt) during 6 MWT. It will be assessed at baseline, 4 th week, 8th week and at 12th week.
Modified Borg Dyspnoea Scale | 12 week
  Changes from baseline will be measured, It is most commonly used to assess symptoms of breathlessness. It starts at number 0 where your breathing is causing you no difficulty at all and progresses through to number 10 where your breathing difficulty is maximal. It will be assess while participants doing 6 MWT.
Fatigue Severity Scale (FSS) | 12 week
  Changes from the baseline Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue on you. The FSS is a short questionnaire that requires you to rate your level of fatigue. The FSS questionnaire contains nine statements that rate the severity of your fatigue symptoms. It will be assess while participants doing 6 MWT.
Adverse events | 12 week
  The number of adverse events resulting from the intervention will be noted.
Change in medication | 12 week
  Any reporting on hospitalization, visits to cardiologist/medical specialist and any change in medication will be recorded on questionnaire.
Adherence to the program | 12 week
  proportion % of the 36 potential sessions of adherent patients will be estimated in each of the periods followed.
Satisfaction score | 12 week
  Patient Assessment of Chronic Illness Care (PACIC) is a psychometrically validated scale, which could serve as a useful tool to assess patient satisfaction with Cardiac Rehabilitation. It is a 22-item self-measurement of how well patients perceive their chronic condition(s) are being managed by their health care team. Patients answer using a Likert scale of answers ranging from 1-5, with 1 signifying "None of the time" and 5 signifying "Always". the overall PACIC score is calculated by averaging scores across all 20 items. Higher scores denote greater satisfaction.
Thigh circumference | 12 week
  Changes will be measured at baseline, 6th week and at 12th week. Thigh circumference (TC) will be measured using a tape measure in centimeter at the mid-trochanterion tibiale lateral site perpendicular to the longitudinal axis while the subject was standing.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Principal Investigator — Riphah International University; Arshad Nawaz Malik, PhD, Study Chair — Riphah International University; Shane Patman, PhD, Study Chair — University of Notre Dame Australia
Locations (2):
- Pakistan (2):
  - Pakistan Railway Hospital, Rawalpindi, Punjab Province
  - Rawalpindi Institute of Cardiology, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No